CLINICAL TRIAL: NCT03563820
Title: Intervention to Improve Resilience and Mental Health in Veterans With Injury, Illness, and/or Disability
Brief Title: Resilience and Well-Being Pilot Study
Status: Completed | Type: Observational
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rhonda Williams, PhD, Attending Psychologist, VA Puget Sound Health Care System
Other Study IDs: 01620
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain; Depression; PTSD; Injuries; Illness, Chronic; Physical Disability
Keywords: Positive Psychology; Resilience; Well-Being
MeSH Terms: conditions — Chronic Pain; Depression; Stress Disorders, Post-Traumatic; Wounds and Injuries; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Resilience and Well-Being Program — The Resilience and Well-Being Program is offered through VA Puget Sound Rehabilitation Care Services as part of standard clinical care offerings. The program includes five (5) positive psychology group sessions once a week for five weeks. Participants will use strengths-based strategies, narrative strategies, and prospective strategies to learn ways to deal with stressful life challenges and improve their mental health and well-being.
  Each participant will be given a brief rating sheet at the end of each session to fill out. The rating sheet will ask participants to rate different aspects of the session (e.g., how helpful or interesting the session was to the participant), if home practice activities were assigned, whether the participant completed the home practice assignment, as well as feedback to improve that session.

SUMMARY:
It is common for Veterans with injuries, illnesses, or physical disabilities to experience depression, post-traumatic stress disorder (PTSD), chronic pain, and other concerns. They may also have goals like becoming happier or better able to cope with challenges that life brings. The purpose of this research study is to learn whether Veterans like and benefit from a 5-week, group-based positive psychology program aimed at improving mental health, resilience, well-being, and quality of life. Participants will be asked to complete several assessments (surveys/interviews) over the course of the study that are not considered part of standard care. Additionally, participants will be asked to participate in a focus group at the end of the study to provide feedback about their experiences in the group.

DETAILED DESCRIPTION:
To participate in this study, Veterans must first be enrolled in the Resilience and Well-Being Program, a 5-week, group-based positive psychology program held at VA Puget Sound as part of standard care. After enrollment, Veterans may choose to enroll in this research study which evaluates the effectiveness of, and satisfaction with, the Resilience and Well-Being Program.

This research study includes two study visits at VA Puget Sound and three assessments over the phone.

Informed Consent Process

This process will take place at the VA Puget Sound. A research staff member will review the details of the study with the participant and answer any questions s/he may have to see if they are interested in participating.

Assessments

1. Baseline Assessment: A research staff member will ask the participant a number of standard questions. The most straightforward of these questions will ask about age, gender, race, ethnicity, education level, employment status, marital status, and military service. Participants will also be asked questions about their medical and mental health treatment use, and any other health problems they may experience. Participants will also be asked questions about potentially stressful life experiences.
2. Post-Group Satisfaction Survey: This survey will happen following the completion of the 5-week group as long as a participant has attended at least one session. Participants will be asked to complete this survey in-person at the end of Session 5. In this survey, participants will be asked questions about how satisfying, engaging, and helpful they thought the program was; what they thought about the program, and whether they experienced any negative effects from participating in the program.
3. Telephone Assessments: Throughout participation in the study, participants will be asked to complete three telephone assessments. Within each assessment, participants will be asked questions relating to:

   * How the participant is feeling
   * Satisfaction with life and well-being
   * Positive and negative emotions
   * Participation and satisfaction with social activities
   * Problems related to very stressful experiences
   * Physical pain and how it is affecting the participant's life
   * Current and past mental health treatment use
   * How likely the participant is to seek mental health treatment
   * Changes in medications, psychological treatment, or new major life events
   * How illness/injury has impacted the participant's life
   * Whether the participant noticed any changes in their life after the group (once the group is over)

The three telephone assessments will occur at the following stages of the study:

* Pre-Group Assessment must be completed before the first group session.
* Post-Group Assessment will occur at the end of the 5-week group period.
* 5-Week Follow-Up Assessment will occur about 5 weeks after the end of the 5-week group period.

Focus Group (Optional)

Participants will be invited to complete a focus group that will last about 60-90 minutes six to eight weeks after the completion of the group to talk about their experiences and satisfaction with the program. Completing the focus group is optional, but encouraged, as researchers would like to receive participant feedback through open discussion to better improve this program for other Veterans. The focus group leaders will use prepared questions to help guide the flow of discussion.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran status (defined as prior service in the US Armed Forces and eligible to receive health care services through Veterans Health Affairs)
2. 18 years of age or older
3. Enrolled, or eligible and willing to enroll, in the Resilience and Well-Being group treatment program (offered as part of standard clinical care in VA Puget Sound Rehabilitation Care Services)
4. Able to read, speak, and understand English
5. Has been seen at least once in the past 12 months in a VAPSHCS clinic that provides rehabilitation services to individuals with rehabilitation needs related to conditions including (but not limited to) multiple sclerosis (MS), traumatic brain injury (TBI), amyotrophic lateral sclerosis (ALS), spinal cord injury (SCI), stroke, myocardial infarction, limb loss, polytrauma, neuromuscular conditions, musculoskeletal problems, impairing but medically unexplained symptoms, and/or pain, OR has a diagnosis of such a condition
6. Positive screen for depression, PTSD, or chronic pain

Exclusion Criteria:

1. Primary psychotic or major thought disorder as listed in participant's medical record or self-reported
2. Psychiatric or behavioral conditions in which symptoms were unstable or severe (e.g., current delirium, mania, psychosis, suicidal ideation, homicidal ideation, active substance use disorder, psychiatric hospitalization) as listed in participant's medical record or self-reported within the past six months
3. Any behavioral, cognitive, or psychiatric issues that would indicate the participant may be inappropriate in a group setting or for this particular group-format intervention, subject to clinician discretion
4. Difficulties or limitations communicating over the telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be Veterans enrolled in the VA Puget Sound Resilience and Well-Being Program, which is offered through VA Puget Sound Rehabilitation Care Services as part of standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Change in Depression from Pre-Group to 5-Weeks Post-Group | Pre-Group (up to 2-weeks prior to Session 1 of group program), Post-Group (immediately after Session 5 of group program, window open up to 4 weeks after), 5-Week Follow-Up (5 weeks after Session 5 of program, window open up to 4 weeks after)
  Change in depression will be measured using the PROMIS Depression Short Form-8A. Responses from each item will be summed to form a total raw score ranging from 8-40. Higher scores indicate higher self-reported levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Williams, Ph.D., Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03563820/ICF_000.pdf